CLINICAL TRIAL: NCT00528021
Title: A Study Evaluating the Safety and Efficacy of BGC20-0582 Lice Treatment Gel for Head Lice Infestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCG20-0582-001
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2010-12-28 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Pediculus Humanus Capitis; Head Lice
Keywords: Head Lice; Lice Infestation; Pediculosis; Pediculosis Capitis
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Subjects are treated either once (day1) or twice (day 1 and 7) with either placebo or 2.5% BGC20-0582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
  Interventions: Drug: BGC20-0582
- 2 (Active Comparator): Subjects are treated either once (day1) or twice (day 1 and 7) with either placebo or 10% BGC20-0582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
  Interventions: Drug: BGC20-0582
- 3 (Active Comparator): Subjects are treated either once (day1) or twice (day 1 and 7) with either placebo or 12.5% BGC20-0582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
  Interventions: Drug: BGC20-0582
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Vehicle Only
  Arms: 4
Drug: BGC20-0582 — BGC20-0582 is a topical gel formulation of a naturally derived product. Subjects are treated either once (day 1) or twice (day 1 and 7) with either placebo or BGC20-0582 at one of the three concentrations. Following application of the BGC20-0582 lice treatment gel of placebo the product is rinsed from the subjects hair.
  Arms: 1; 2; 3

SUMMARY:
The main purpose of this study is to investigate the safety and efficacy of an investigational treatment for head lice infestation against a placebo.

DETAILED DESCRIPTION:
The main purpose of this study is to investigate the safety and efficacy of an investigational treatment for head lice infestation against a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. The subject and/or his/her parent/legal guardian have provided written informed consent, and, if appropriate, the child has provided assent.
2. Male or female subjects who are between the ages of 2 years (24 months) and 70 years old when consent is signed.
3. Infestation with head lice as demonstrated by the presence of live lice prior to first treatment.
4. Willing and able to attend all study visits as scheduled.
5. Females of childbearing potential must have a negative urine pregnancy test at screening and before receiving a second treatment, if necessary.

Exclusion Criteria:

1. Subject and/or legal guardian has not signed informed consent.
2. Subject was treated for pediculosis within 2 weeks prior to the screening evaluation.
3. Subject with an infestation of body lice or pubic lice.
4. Subject is suffering from a condition likely to require medical attention, including administration of oral or systemic antibiotics, oral or systemic corticosteroids, or any other treatment, which in the opinion of the investigator and visiting physician could influence the results of the study.
5. Subject with other diagnoses which, in the opinion of the investigator, would interfere with efficacy or safety assessments or would preclude study participation.
6. Subject with very short (shaved) hair.
7. Subject who will not be available for follow up visits.
8. Subject has been treated with a systemic antibiotic within the previous two weeks before screening.
9. Subject has been previously enrolled in any clinical study within the past 30 days; subject may not participate in another study while participating in this study.
10. Subject with history of allergy/sensitivity to active ingredient or related products; or any ingredients commonly included in hair products such as shampoos, hair conditioners, or styling aids.
11. Pregnant and/or nursing females.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Global Health Associates of Miami Inc, Florida City, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.5% BGC20-0582: Active Comparator: 1
  Subjects are treated either once (day 1) or twice (day 1 and 7) with either placebo or 2.5% BGC20-0582 topically. Following application of the BG20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
- 10% BGC20-0582: Active Comparator: 2
  Subjects are treated either once (day 1) or twice (day 1 and 7) with either placebo or 10% BGC20-0582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
- 12.5% BGC20-0582: Active Comparator: 3
  Subjects are treated either once (day 1) or twice (day 1 and 7) with either placebo or 12.5% BGC20-0582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
- Vehicle: Placebo Comparator: 4
Period: Overall Study
Arm/Group | 2.5% BGC20-0582 | 10% BGC20-0582 | 12.5% BGC20-0582 | Vehicle
Started | 59 | 59 | 56 | 56
Completed | 42 | 46 | 49 | 47
Not Completed | 17 | 13 | 7 | 9
Not completed — Lack of Efficacy | 17 | 13 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5% BGC20-0582 | 10% BGC20-0582 | 12.5% BGC20-0582 | Vehicle | Total
Number analyzed (Participants) | 59 | 59 | 56 | 56 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 56 | 55 | 55 | 221
  Between 18 and 65 years | 4 | 3 | 1 | 1 | 9
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (11.5) | 13.5 (12.1) | 13 (10.2) | 12.3 (8.8) | 12.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 49 | 49 | 206
  Male | 5 | 5 | 7 | 7 | 24
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 56 | 56 | 230

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure
Description: Count of participants with No live lice
Time Frame: Day 15 or 22
Measure: Count of Participants; unit: Participants
Groups:
- 2.5% BGC20-0582: Active Comparator: 1
  Subjects are treated either once (day 1) or twice (day 1 and 7) with either placebo or 2.% BGC20-582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
- 10% BGC20-0582: Active Comparator: 2
  Subject's are treated either once (day 1) or twice (day 1 and 7) with either placebo or 10% BGC20-0582 topically. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
- 12.5% BGC20-0582: Active Comparator: 3
  Subject's are treated either once (day 1) or twice (day 1 and 7) with either placebo or 12.5% BG20-0582 TOPICALLY. Following application of the BGC20-0582 lice treatment gel or placebo, the product is rinsed from the subject's hair.
Arm/Group | 2.5% BGC20-0582 | 10% BGC20-0582 | 12.5% BGC20-0582 | Vehicle
Number analyzed (Participants) | 42 | 46 | 49 | 47
Participants | 30 | 28 | 35 | 32

ADVERSE EVENTS:
Arm/Group | 2.5% BGC20-0582 | 10% BGC20-0582 | 12.5% BGC20-0582 | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 13/59 | 10/59 | 16/56 | 11/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5% BGC20-0582 (N=59) | 10% BGC20-0582 (N=59) | 12.5% BGC20-0582 (N=56) | Vehicle (N=56)
Application site irritation (General disorders) | 8 (8) | 5 (5) | 8 (8) | 3 (3)
Application site pruritis (General disorders) | 4 (4) | 2 (2) | 2 (2) | 5 (5)
Dandruff (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less